CLINICAL TRIAL: NCT02191111
Title: A Cluster-randomized Controlled Knowledge Translation Feasibility Study in Alberta Community Pharmacies Using the PARiHS Framework
Brief Title: A Cluster-randomized Controlled Knowledge Translation Feasibility Study in Alberta Community Pharmacies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); University of Waterloo (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00047475; 201300643 (Other Grant/Funding Number: Alberta Innovates - Health Solutions)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2018-05

CONDITIONS: Chronic Diseases
Keywords: Pharmacist; Pharmacy practice; Patient care; Community pharmacy; Hypertension; Diabetes; Dyslipidemia; Pharmaceutical care
MeSH Terms: conditions — Chronic Disease; Hypertension; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Task-focused facilitation (Experimental): An external, task-focused facilitation, informed by an evaluation of contextual factors using the Alberta Context Tool (ACT), will be applied to train community pharmacies to develop alternative team processes that enable a greater number of medication management services to be provided to patients with diabetes, hypertension, and/or dyslipidemia.
  Interventions: Behavioral: Task-focused facilitation
- Control (No Intervention): These sites will continue practice as usual, with no contact from study staff.

INTERVENTIONS:
Behavioral: Task-focused facilitation — An external, task-focused facilitation, informed by an evaluation of contextual factors using the Alberta Context Tool (ACT), will be applied to train community pharmacies to develop alternative team processes that enable a greater number of medication management services to be provided to patients with diabetes, hypertension, and/or dyslipidemia.
  Arms: Task-focused facilitation

SUMMARY:
Background: Despite evidence of benefit for pharmacist involvement in chronic disease management, the provision of these services in community pharmacy has been suboptimal. The Promoting Action on Research Implementation in Health Services (PARiHS) framework suggests that for knowledge translation to be effective, there must be evidence of benefit, a context conducive to implementation, and facilitation to support uptake. We hypothesize that while the evidence and context components of this framework are satisfied, that uptake into practice has been insufficient because of a lack of facilitation. This protocol describes the rationale and methods of a feasibility study to test a facilitated pharmacy practice intervention based on the PARiHS framework, to assist community pharmacists in increasing the number of formal and documented medication management services completed for patients with diabetes, dyslipidemia, and hypertension.

Methods: A cluster-randomized before-after design will compare ten pharmacies from within a single organization, with the unit of randomization being the pharmacy. Pharmacies will be randomized to facilitated intervention based on the PARiHS framework or usual practice. The Alberta Context Tool will be used to establish the context of practice in each pharmacy. Pharmacies randomized to the intervention will receive task-focused facilitation from an external facilitator, with the goal of developing alternative team processes to allow the greater provision of medication management services for patients with diabetes, hypertension, and dyslipidemia. The primary outcome will be a process evaluation of the needs of community pharmacies to provide more clinical services, the acceptability and uptake of modifications made, and the willingness of pharmacies to participate. Secondary outcomes will include the change in the number of formal and documented medication management services in the aforementioned chronic conditions provided 6 months before, versus after, the intervention between the two groups, and identification of feasible quantitative outcomes for evaluating the effect of the intervention on patient care outcomes.

Results: To date, the study has identified and enrolled the ten pharmacies required and initiated the intervention process.

Conclusion: This study will be the first to examine the role of facilitation in pharmacy practice, with the goal of scalable and sustainable practice change.

DETAILED DESCRIPTION:
Please see the following publication for a detailed description of the work:

Pilot and Feasibility Studies 01/2015; 1(2). DOI: 10.1186/2055-5784-1-2

ELIGIBILITY:
Inclusion Criteria:

* Pharmacies: Community pharmacy locations of a medium-sized pharmacy chain with an interest in and the ability to provide medication management services, but have not fully integrated these activities
* Patients: Any Alberta residents qualifying for pharmacy clinical services as defined by the Alberta Pharmacy Fee Framework

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross T Tsuyuki, PharmD, MSc, Principal Investigator — University of Alberta; Meagen M Rosenthal, BA, MA, PhD, Study Director — University of Alberta; Sherilyn KD Houle, BSP, PhD, Study Director — University of Waterloo
Locations (1):
- EPICORE Centre, University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Rosenthal MM, Tsuyuki RT, Houle SK. A cluster-randomized controlled knowledge translation feasibility study in Alberta community pharmacies using the PARiHS framework: study protocol. Pilot Feasibility Stud. 2015 Jan 12;1:2. doi: 10.1186/2055-5784-1-2. eCollection 2015. PMID 27965782
- [Derived] Houle SK, Charrois TL, Faruquee CF, Tsuyuki RT, Rosenthal MM. A randomized controlled study of practice facilitation to improve the provision of medication management services in Alberta community pharmacies. Res Social Adm Pharm. 2017 Mar-Apr;13(2):339-348. doi: 10.1016/j.sapharm.2016.02.013. Epub 2016 Mar 8. PMID 27017157
- See also: Study protocol — http://www.pilotfeasibilitystudies.com/content/1/1/2

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: pharmacies
Period: Overall Study
Arm/Group | Task-focused Facilitation | Control
Started | NA; 5 pharmacies (Number of participants assigned NA because the unit of analysis was pharmacies not patients.) | NA; 5 pharmacies (Number of participants assigned NA because the unit of analysis was pharmacies not patients.)
Completed | NA; 5 pharmacies (Number of participants assigned NA because the unit of analysis was pharmacies not patients.) | NA; 5 pharmacies (Number of participants assigned NA because the unit of analysis was pharmacies not patients.)
Not Completed | NA; 0 pharmacies | NA; 0 pharmacies

BASELINE CHARACTERISTICS:
Population: Unit of analysis pharmacies
Units Other Than Participants: Pharmacies
Groups:
- Total: Total of all reporting groups
Arm/Group | Task-focused Facilitation | Control | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Pharmacies) | 5 | 5 | 10
Age, Customized [Number; unit: Age data not collected]
  Pharmacies | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Pharmacies]
  Pharmacies | 0 | 0 | 0
Alberta context tool, semi-structured interviews, medication management counts, close out interviews [Mean (Full Range); unit: units on a scale] — The Alberta Context Tool is designed to obtain a measure of the organizational culture of a clinical setting. The scale is measured on a series of 5-point Likert scales from strongly disagree to strongly agree or never to almost always. Each of the five items is assigned a number from 1 (strongly disagree/never) to 5 (strongly agree/almost always). Composite scores (mean scores taken of responses to each item) are calculate for each of the sub-scales and combined for a total score. The higher the score the more a site demonstrates the sub-scale characteristic.
  units on a scale | 2.86 [1 to 5] | 3.14 [1 to 5] | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Change in Service Counts From Baseline to End of Intervention Period
Description: Difference in the number of billable services (influenza vaccinations, Comprehensive Annual Care Plans and follow-ups, and Standard Medication Management Assessments and follow-ups) between the intervention period and the 6-months prior to intervention (baseline)
Time Frame: 6 month intervention period vs. 6 month baseline prior to intervention
Population: Units of measure were community pharmacies
Measure: Count of Units; unit: Billable pharmacy services
Units Other Than Participants: Billable pharmacy services
Arm/Group | Task-focused Facilitation | Control
Number analyzed (Participants) | 5 | 5
Number analyzed (Billable pharmacy services) | 4557 | 5886
Billable pharmacy services
  CACP (Baseline) | 172 | 284
  CACP (Study Period) | 121 | 166
  CACP Follow-Up (Baseline) | 295 | 507
  CACP Follow-Up (Study Period) | 106 | 372
  SMMA (Baseline) | 50 | 115
  SMMA (Study Period) | 46 | 64
  SMMA Follow-Up (Baseline) | 67 | 105
  SMMA Follow-Up (Study Period) | 41 | 88
  SMMA Diabetes (Baseline) | 3 | 4
  SMMA Diabetes (Study Period) | 1 | 1
  SMMA Diabetes Follow-Up (Baseline) | 8 | 5
  SMMA Diabetes Follow-Up (Study Period) | 4 | 5
  SMMA Tobacco (Baseline) | 21 | 6
  SMMA Tobacco (Study Period) | 8 | 12
  SMMA Tobacco Follow-Up (Baseline) | 4 | 4
  SMMA Tobacco Follow-Up (Study Period) | 5 | 6
  Influenza Vaccinations (Baseline) | 406 | 2
  Influenza Vaccinations (Study Period) | 3199 | 4140

ADVERSE EVENTS:
Description: Adverse events were not collected.
Arm/Group | Task-focused Facilitation | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No